CLINICAL TRIAL: NCT01376843
Title: Conversion Rate of TST and Quantiferon-TB Gold In Tube Assay in Health Care Workers
Brief Title: Conversion Rate of (TST) Tuberculin Skin Test and Quantiferon-TB Gold In Tube Assay in Health Care Workers
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0161
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Tuberculosis
Keywords: latent tuberculosis in health care workers
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood for perfoming Quantiferon-TB Gold in tube assay
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Health care workers: health care workers who performed TST or Quantiferon-TB Gold In tube assay before

SUMMARY:
The purpose of this study is to access conversion rate of TST (Tuberculin skin test) and Quantiferon-TB Gold In tube assay in health care workers.

ELIGIBILITY:
Inclusion Criteria:

* age 20-75, men and women
* participant who was enrolled in the study of latent tuberculosis in health care worker (IRB No.4-2009-0187)
* high risk or low risk health care worker who was performed TST or Quantiferon-TB Gold In tube assay before

Exclusion Criteria:

* age < 20
* person who don't agree with enrollment
* illiterate
* person who is diagnosed as active tuberculosis now
* person who has history of hypersensitivity on PPD (tuberculin purified protein derivative)
* pregnant woman
* person who is treated as active tuberculosis

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: health care workers who performed TST or Quantiferon-TB Gold In tube assay before
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
conversion rate of latent tuberculosis infection in hospital workers | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Menzies D, Fanning A, Yuan L, Fitzgerald M. Tuberculosis among health care workers. N Engl J Med. 1995 Jan 12;332(2):92-8. doi: 10.1056/NEJM199501123320206. No abstract available. PMID 7990907
- [Background] Jiamjarasrangsi W, Hirunsuthikul N, Kamolratanakul P. Tuberculosis among health care workers at King Chulalongkorn Memorial Hospital, 1988-2002. Int J Tuberc Lung Dis. 2005 Nov;9(11):1253-8. PMID 16333934
- [Background] Schwartzman K, Loo V, Pasztor J, Menzies D. Tuberculosis infection among health care workers in Montreal. Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):1006-12. doi: 10.1164/ajrccm.154.4.8887599.
- [Background] Kruuner A, Danilovitsh M, Pehme L, Laisaar T, Hoffner SE, Katila ML. Tuberculosis as an occupational hazard for health care workers in Estonia. Int J Tuberc Lung Dis. 2001 Feb;5(2):170-6. PMID 11258511